CLINICAL TRIAL: NCT06111443
Title: Effect of Dapagliflozin on the Recurrence of Atrial Tachyarrhythmia in Patients Undergoing Catheter Ablation of Atrial Fibrillation - A Randomized Open-Label Phase III Trial
Brief Title: Effect of Dapagliflozin on the Recurrence of Atrial Tachyarrhythmia in Patients Undergoing Catheter Ablation of Atrial Fibrillation
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPRPG8N0011
Record Dates: First submitted 2023-08-31; First posted 2023-11-01 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-08

CONDITIONS: Atrial Fibrillation Recurrent; Catheter Ablation
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin (FORXIGA) 10 mg QD for 3 months
  Interventions: Drug: Dapagliflozin 10 mg [Farxiga]
- Usual care (No Intervention): guideline-direct usual care

INTERVENTIONS:
Drug: Dapagliflozin 10 mg [Farxiga] — Dapagliflozin 10 mg [Farxiga] for 3 months after catheter ablation of atrial fibrillation
  Arms: Dapagliflozin

SUMMARY:
The goal of this clinical trial is to test the effect of Dapagliflozin on the Recurrence of Atrial Tachyarrhythmia in Patients Undergoing Catheter Ablation of Atrial Fibrillation. The main questions it aims to answer are:

• If Dapagliflozin will reduce the recurrence of all atrial tachyarrhythmias [atrial fibrillation (AF), atrial flutter (AFL) and atrial tachycardia (AT)] greater than 30 seconds during one-year follow-up after catheter ablation.

Participants will receive Dapagliflozin (FORXIGA) 10 milligram (mg) once a day (QD) for 3 months after catheter ablation of atrial fibrillation. Researchers will compare patients who receive usual care to see if Dapagliflozin will reduce the recurrence of all atrial tachyarrhythmias (AF/AFL/AT) during one-year follow-up after catheter ablation.

DETAILED DESCRIPTION:
This trial is the third phase of random allocation and non-blind trial. It is divided into study group and control group. The study group is Dapagliflozin therapy, and the treatment period is three months post catheter ablation. The control group is usual care (without Dapagliflozin). The follow-up observation period will be one year after catheter ablation. This trial was performed at Kaohsiung Chang Gung Memorial Hospital and Chang Gung Memorial Hospital, Linkou, and Chiayi branches, and it is a multi-center trial. The study flow chart is as follows.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give written informed consent
* Men and women age >= 20 years.
* Paroxysmal, persistent or long-standing persistent atrial fibrillation
* eGFR >= 25 ml/min/1.73 m2

Exclusion Criteria:

* Receiving therapy with a sodium-glucose cotransporter 2 (SGLT2) inhibitor prior to randomization, or intolerance to an SGLT2 inhibitor.
* Type 1 diabetes mellitus
* Acute coronary syndrome, coronary revascularization (percutaneous coronary intervention or Coronary artery bypass grafting), ablation of atrial flutter/fibrillation, ischemic stroke, and transient ischemic attack within 12 weeks prior to randomization
* Active malignancy
* Women of child-bearing potential who have a positive pregnancy test at randomization or who are breast-feeding
* A life expectancy of fewer than 2 years due to any non-cardiovascular condition, based on the investigator's clinical judgment
* Expected surgery for structural heart disease, and secondary atrial fibrillation (due to cardiac surgery, infection, or hyperthyroidism)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Freedom from all atrial tachyarrhythmias (AF/AFL/AT) | 3,6 and 12 months after ablation
  Freedom from all atrial tachyarrhythmias (AF/AFL/AT) greater than 30 seconds (as documented by 7-day Holter test at 3, 6, and 12-month follow-up) and 12-lead electrocardiogram (ECG) performed at cardiovascular (CV) outpatient department (OPD) follow-up within one-year post catheter ablation. (unit: %)

SECONDARY OUTCOMES:
Freedom from all atrial tachyarrhythmias (AF/AFL/AT) excluding the 3-month blanking period | 6 and12 months after ablation
  Freedom from all atrial tachyarrhythmias (AF/AFL/AT) greater than 30 seconds (as documented by 7-day Holter at 6 and 12-month follow-up) and 12-lead ECG performed at CV OPD follow-up since 3 months post catheter ablation within one year post catheter ablation. (a conventional 3-month blanking period from catheter ablation was used in both groups during which arrhythmia recurrences were not counted toward the recurrent endpoint) (unit: %)
Freedom from all atrial tachyarrhythmias (AF/AFL/AT) within 3-month blanking period | 3 months after ablation
  Freedom from all atrial tachyarrhythmias (AF/AFL/AT) greater than 30 seconds (as documented by 7-day Holter at 3-month follow-up) or 12-leads ECG within 3 months following index ablation (within blanking period) (unit: %)
Total mortality or hospitalization due to CV cause | 12 months after ablation
  Total mortality or hospitalization due to cardiovascular cause within one year after ablation (unit: %)
Left atrial (LA) size (LA dimension and LA volume index) by echocardiography | 6 and 12 months
  Left atrial (LA) size (LA dimension in mm and LA volume index in mL/m2) by echocardiography at 6 and 12 months
AF quality of life (QOL) by AF Effect On Quality-Of-Life (AFEQT) questionnaire score | 1,3,6,9 and 12 months
  Change in AF QOL at 1 month, 3 months, 6 months, 9 months and 12 months after receiving catheter ablation relative to baseline: defined as a change in AF QOL assessed in the validated AFEQT questionnaire score. (no unit)
N-terminal pro-brain natriuretic peptide (NT-proBNP) level | 3 and 12 months
  Blood test for plasma NT-proBNP level in pg/ml
Glycated Hemoglobin (HBA1c) | 3 and 12 months
  HBA1c in %, serum creatinine in mg/dl
Creatinine (Cr) and estimated Glomerular filtration rate (eGFR) | 3 and 12 months
  serum Cr in mg/dl, estimated Glomerular filtration rate (eGFR) by MDRD formula in ml/min per 1.73 m2 (calculated according to serum Cr, age, and sex)
Urine albumin/Cr ratio level | 3 and 12 months
  Urine albumin/Cr ratio in mg/g
Repeated catheter ablation or cardioversion for atrial tachyarrhythmia | 12 months
  Repeated catheter ablation or cardioversion for atrial tachyarrhythmia within one year (unit: %)
Adverse events: hypoglycemia, hypotension, hypokalemia, renal function deterioration | 12 months
  Adverse events: hypoglycemia, hypotension, hypokalemia, renal function deterioration (defined as decline in the estimated GFR of at least 50%) (unit:%)
AF burden | 3,6 and 12 months
  AF burden in % documented by 7-day Holter at 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Lung Chen, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kaoshiung Chang Gung Memorial, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided